CLINICAL TRIAL: NCT03619681
Title: A Single Arm, Open Lable, Dose Escalation Phase I Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Preliminary Efficacy of KN026 Monotherapy in Patients With HER2-positive Advanced Malignant Breast and Gastric Cancer
Brief Title: Trial of KN026 in Patients With HER2-positive Advanced Malignant Breast Cancer and Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN026-CHN-001
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Gastric Cancer
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN026 (Experimental)
  Interventions: Drug: KN026

INTERVENTIONS:
Drug: KN026 — Patient will be intravenously administrated with one dose of KN026. dosing interval may be adjusted during the study based on emerging data from this trial and/or from other trial.

SUMMARY:
This is a first-in-human (FIH), open-label, phase 1 dose-escalation study of KN026 in subjects with HER2 positive advanced breast and Gastric Cancer. The standard "3 + 3" design was used for dose escalation. There are 5 proposed dose levels which are 5, 10, 15, 20 and 30 mg/kg, but dosing interval may be adjusted during the study (such as QW, OR Q2W, OR Q3W) based on emerging data from this trial and/or from phase 1 trial of KN026 in other country. Dose escalation will continue until the maximum tolerated dose (MTD) is reached or if MTD is not found, dose escalation will continue until the MAD of 20 mg / kg is reached. Dose expansion will carried out in 20 mg/kg Q2W and 30 mg/kg Q3W.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject >= 18 years and =<75 years.
* Histologically or cytologically confirmed, locally advanced unresectable or metastatic breast cancer or gastric cancer.
* ECOG score 0 or 1.
* Life expectancy >3 months.
* According to the definition of RECIST1.1, the patient has at least one measurable lesion.
* Adequate organ function prior to start treatment with KN026.
* Able to understand, voluntarily participate and willing to sign the ICF.
* Subjects (women of child-bearing potential and males with fertile female partner) must be willing to use viable contraception method.

Exclusion Criteria:

* Accepted any other anti-tumor drug therapies within 4 weeks before fist dose.
* Accepted radiotherapy within 4 weeks before enrollment(Subjects are eligible, which accepted palliative therapies within 2 weeks before the first dose of KN026 for osseous metastatic and all the AEs recovered).
* An anthracyclines antibiotic treatment, such as doxorubicin (Adriamycin) was received exceeding 300 mg/m² within 90 days before first KN026 dosing, or other equivalent dose antharcyclines.
* Subjects are eligible with clinically controlled and stable neurologic function >= 4 weeks, which is no evidence of CNS disease progression; Subjects with spinal cord compression and cancerous meningitis are not eligible.
* Pregnant or nursing females；or intend pregnancy within this study period or within 6 monthes after the end of this study.
* Has not recovered (ie, >Grade 1) from AEs except alopecia and anemia.
* History of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.
* Severe chronic and active infection, need to system antibiosis/antiviral treatment.
* Cavity effusion (pleural effusion, ascites, pericardial effusion, etc.) are not well controlled, and need locally treatment or repeated drainage. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
The proportion of patients experiencing dose limiting toxicities. | From screening to up to 28 days

SECONDARY OUTCOMES:
Percentage of participants with adverse events (AEs), serious adverse events (SAEs) and AEs of special interest. | From screening to up to 112 days
Percentage of participants who experience laboratory abnormalities and/or adverse events as defined by CTCAE that are related to treatment | From screening to up to 112 days
Maximum observed serum concentration (Cmax) of KN026. | Throughout the duration of the study; up to 84 days
Time of Maximum observed serum concentration (Tmax) of KN026. | Throughout the duration of the study; up to 84 days
Adjusted geometric means of area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUC(0-T)) for KN026. | Throughout the duration of the study; up to 84 days
Serum Half-life (T-HALF) of KN026. | Throughout the duration of the study; up to 84 days.
Serum clearance (CL) of KN026. | Throughout the duration of the study; up to 84 days
Volume of distribution at steady state (VSS) of KN026. | Throughout the duration of the study; up to 84 days
Frequency and titer of anti-KN026 antibody. | Throughout the duration of the study; up to 2 years.
The proportion of patients with an objective response (partial response or complete response) as defined by RECIST 1.1 criteria. | Throughout the duration of the study; up to 2 years.
Progression free survival according to RECIST 1.1 criteria. | Throughout the duration of the study; up to 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Hospital, Shanghai, China